CLINICAL TRIAL: NCT06999941
Title: A Prospective Observational Study Evaluating the Efficacy and Safety of Deucravacitinib in the Treatment of Moderate to Severe Plaque Psoriasis Patients With Eczematous Features in a Real-world Research
Brief Title: A Real-world Study of Deucravacitinib in the Treatment of Moderate to Severe Plaque Psoriasis With Eczematous Features
Status: Enrolling by invitation | Type: Observational
Sponsor: Xi Tan (Other)
Responsible Party: Sponsor-Investigator, Xi Tan, physician-in-charge, Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine
Organization: Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine (Other)
Other Study IDs: 20240924103453152
Record Dates: First submitted 2025-05-12; First posted 2025-05-31 (Actual); Last update posted 2025-05-31 (Actual); Status verified 2025-04

CONDITIONS: Psoriasis; Eczema; JAK Inhibitor
MeSH Terms: conditions — Psoriasis; Eczema | interventions — deucravacitinib

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Fresh frozen tissue for RNA-seq and RT-PCR, Formalin fixed tissue for IHC and HE
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: Deucravacitinib 6mg po qd — oral administration

SUMMARY:
Emerging evidence indicates that psoriasis and eczema can coexist in the same patient, with reported co-prevalence rates ranging from 0.17% to 20%, suggesting that these conditions may represent a disease spectrum-referred to as Psoriasis Eczema (PsEma). Moreover, paradoxical eczema has been observed in approximately 1% to 12.1% of psoriasis patients undergoing biologic therapy, with up to 61% of affected individuals discontinuing treatment due to eczematous flares. These findings underscore an urgent need for therapeutic agents that are efficacious for PsEma.

Tyrosine kinase 2 (TYK2), a member of the Janus kinase (JAK) family, is known to mediate critical signaling pathways involved in psoriasis pathogenesis, including those of type I interferons, interleukin (IL)-12, and IL-23. Additionally, TYK2 forms heterodimers with other JAK family members-such as JAK1 or JAK2-to transduce signals from cytokines like IL-13 and IL-22, which are centrally implicated in the pathophysiology of eczema. Based on this molecular profile, we hypothesize that TYK2 inhibition may not only avoid inducing eczematous reactions in psoriasis patients but may also alleviate eczematous inflammation by interfering with JAK1(JAK2)/TYK2-mediated IL-13 and IL-22 signaling.

Deucravacitinib, a selective allosteric TYK2 inhibitor, has shown promising results in our clinical practice, demonstrating improvements in both psoriatic and eczematous manifestations among patients with PsEma. This study aims to prospectively evaluate the efficacy and safety of deucravacitinib in PsEma patients over a 16-week treatment period. In parallel, transcriptomic profiling of peripheral blood and lesional skin will be performed to elucidate the immunological landscape and molecular signatures underlying PsEma, thereby contributing valuable clinical and mechanistic insights into its diagnosis and management.

DETAILED DESCRIPTION:
Eczema-like psoriasis, also referred to as psoriasis-eczema overlap, is a distinct clinical and immunopathological entity that presents with features of both chronic plaque psoriasis and atopic dermatitis (AD). It is increasingly recognized in dermatological practice but remains under-characterized in the literature. Clinically, patients may exhibit erythematous, scaly plaques typical of psoriasis, alongside intense pruritus, oozing, and lichenification more typical of eczematous dermatitis. Histologically, such lesions often display psoriasiform epidermal hyperplasia with superimposed spongiosis, eosinophilic infiltration, and crusting-hallmarks of an eczematous response.

ELIGIBILITY:
Inclusion Criteria:

1.patients who present typical psoriasis and typical eczema; 2.patients present untypical psoriasis lesions, biopsy result reveals both psoriasis and eczema features; 3.BSA≥3 and IGA≥3.

Exclusion Criteria:① Local use of therapeutic drugs (such as glucocorticoids, calcineurin inhibitors, etc.) within 2 weeks Vitamin D derivatives, retinoid drugs); Received biological treatment within 4 weeks or 4 half lives Agents or their immunosuppressive/immunomodulatory agents (such as cyclosporine, methotrexate, JAK inhibitors);

* Suffering from active autoimmune diseases; Active tuberculosis infection; Hepatitis B surface antigen positive; Uncontrolled systemic diseases such as heart failure, cerebrovascular disease, and liver and kidney dysfunction;

  * Known or suspected history of immunosuppression, or although the infection has disappeared, it has been assessed by the researcher as possible Frequent publication of authors;

    * History of malignant tumors in the past, or current occurrence of any malignant tumors (excluding basal tumors cured for ≥ 1 year) Cell carcinoma, local squamous cell carcinoma of the skin, or cervical cancer in situ;

      * Pregnant or lactating women, or those with pregnancy plans during the trial period.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: clinical patients
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2025-04-24 (Actual); Primary Completion 2026-08-30 (Estimated); Study Completion 2026-08-30 (Estimated)

PRIMARY OUTCOMES:
Percentage of patients with PASI75 | From enrollment to the end of treatment at 16 weeks
Change from baseline in PASI | From enrollment to the end of treatment at 16 weeks
Proportion of patients with s-PGA 0 or 1 | From enrollment to the end of treatment at 16 weeks

SECONDARY OUTCOMES:
Proportion of patients with IGA 0 or 1 | From enrollment to the end of treatment at 16 weeks
change of BSA in eczema from baseline | From enrollment to the end of treatment at 16 weeks
Changes from baseline in WI-NRS | From enrollment to the end of treatment at 16 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai general hospital, Shanghai Jiao Tong University School of Medicine, Shanghai, Shanghai Municipality, China